CLINICAL TRIAL: NCT06471101
Title: Applying Artificial Intelligence to Identify Subphenotypes of Acute Kidney Injury in Mexican Patients With Severe COVID-19
Acronym: IA-COVAKI
Status: Completed | Type: Observational
Sponsor: Instituto Nacional de Enfermedades Respiratorias (Other Government)
Responsible Party: Principal Investigator, Elizabeth Santiago Del Angel, Ph D. in computer science, Instituto Nacional de Enfermedades Respiratorias
Other Study IDs: C38-23
Record Dates: First submitted 2024-06-18; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: COVID-19; Acute Kidney Injury
Keywords: machine learning; artificial intelligence
MeSH Terms: conditions — COVID-19; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: clusters — clustering

SUMMARY:
The goal of this observational study was to identify subphenotypes of acute kidney injury patients with COVID-19, and the investigators analyzed their impact on mortality. The study included demographic and clinical variables of the participants. The implementation of Machine Learning algorithms and Artificial Intelligence methods are used, and some specific implementations were designed for the analysis, where each group was characterized by traditional statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 15 years old, hospitalized, and with severe acute respiratory syndrome (SARS-CoV-2) positive confirmation.

Exclusion Criteria:

* Patients who did not have at least 1 creatinine measurement.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with acute kidney injury and COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 2934 (Actual)
Dates: Start 2024-06-18 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Subphenotypes of acute kidney injury in patients | Through study completion, an average of one month
  Number of acute kidney injury subphenotypes in patients with COVID-19

SECONDARY OUTCOMES:
Mortality of acute kidney injury patients | Through study completion, an average of one month
  Differences between mortality rates in acute kidney injury subphenotypes of patients with COVID-19
Severity of acute kidney injury patients | Through study completion, an average of one month
  Differences between severity stages in acute kidney injury subphenotypes of patients with COVID-19
Non-recovery in acute kidney injury patients | Through study completion, an average of one month
  Differences between non recovery rates in acute kidney injury subphenotypes of patients with COVID-19
Renal replacement therapy requirement in acute kidney injury patients | Through study completion, an average of one month
  Differences between renal replacement therapy requirement rates in acute kidney injury subphenotypes of patients with COVID-19
Length of stay of acute kidney injury patients | Through study completion, an average of one month
  Differences in-hospital length of stay in acute kidney injury subphenotypes of patients with COVID-19.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Enfermedades Respiratorias, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided